CLINICAL TRIAL: NCT00815386
Title: Safety and Efficacy of Percutaneous Transvenous Mitral Annuloplasty System to Reduce Mitral Valve Regurgitation in Patients With Heart Failure
Brief Title: Safety and Efficacy Study of the PTMA Device to Reduce Mitral Valve Regurgitation in Patients With Heart Failure
Acronym: PTOLEMY2Canada
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Company ended operations in January 2011
Sponsor: Viacor (Industry)
Collaborators: Duke University (Other); Medifacts International Corporation (Industry)
Responsible Party: Katharine M Stohlman, VP Regulatory Affairs, Viacor, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-037P
Record Dates: First submitted 2008-12-26; First posted 2008-12-30 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Mitral Regurgitation; Heart Failure
Keywords: mitral valve; heart failure; mitral regurgitation; annuloplasty; coronary sinus
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTMA implanted (Experimental): Enrolled patients receiving a PTMA implant
  Interventions: Device: Percutaneous transvenous mitral annuloplasty

INTERVENTIONS:
Device: Percutaneous transvenous mitral annuloplasty — Catheterization procedure with anesthesia requiring subclavicular puncture, catheterization of the right atrium and coronary sinus vein, placement and optimization of the PTMA device with access hub remaining subcutaneous at the clavicle.
  Other Names: mitral annuloplasty; sinoplasty

SUMMARY:
Improvement in heart failure with moderate to severe mitral regurgitation using a percutaneously delivered implantable device residing in the coronary sinus

DETAILED DESCRIPTION:
Device under Test: The Viacor® Percutaneous Transvenous Mitral Annuloplasty (PTMA) system comprises a sterile implantable cardiac device and associated custom accessories to assist implantation. The PTMA system is intended to treat functional mitral regurgitation (MR) in a heart failure patient by a less invasive method than surgical annuloplasty with greater relief of symptoms than medical management alone.

Study Objective: Functional mitral regurgitation is associated with an adverse prognosis in the heart failure patient. The objective of this study is to evaluate whether PTMA is effective in reducing mitral regurgitation in heart failure patients and whether this reduction is associated with a moderation in the adverse progression of heart failure symptoms.

Hypothesis under Test: Reduction of the severity of functional mitral regurgitation from baseline, as defined by a composite improvement of quantitative echocardiographic metrics, can be achieved safely with the PTMA device and will be associated with a measurable moderation of adverse progression of heart failure symptoms and a moderation of the deterioration of exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patient has moderate functional MR: regurgitant orifice area >/= 0.20cm2 or regurgitant volume >/= 30 mL/beat or regurgitant fraction >/= 30%
* Symptomatic heart failure NYHA Class II to IV
* LV dysfunction (25% < LVEF < 50% by echocardiography) OR dilated mitral annulus > 30mm

Exclusion Criteria:

* MR of organic origin
* Severe mitral leaflet tethering
* History of MI or PCI within 60 days of study procedure
* Inability to walk a minimum of 100 meters in 6 minutes
* Significant left main stenosis or proximal circumflex stent
* Indication of non-patent CSO or discontinuous CS-GCV-AIV
* Bi-ventricular with leads in CS or other devices impeding device placement
* Severe aortic valvular disease
* Chronic corticosteroid use other than < 20mg prednisone for arthritis
* Significant co-morbidities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of mitral regurgitation | 6 months
Freedom from major adverse cardiac events (death, MI, emergent cardiac surgery, and stroke). | 30 days

SECONDARY OUTCOMES:
Improvement of 6 minute walk distance | 6 months
Improvement in Quality of Life Score | 6 months
Reduction of mitral regurgitation | 6 months
Freedom from procedure-related or device-related major adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luc Bilodeau, MD, Principal Investigator — Montreal Heart Institute
Locations (3):
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Royal Victoria Hospital, McGill University Medical Center, Montreal, Quebec
  - Laval Hospital, Quebec Heart-Lung Institute, Québec, Quebec

REFERENCES:
- [Background] Dubreuil O, Basmadjian A, Ducharme A, Thibault B, Crepeau J, Lam JY, Bilodeau L. Percutaneous mitral valve annuloplasty for ischemic mitral regurgitation: first in man experience with a temporary implant. Catheter Cardiovasc Interv. 2007 Jun 1;69(7):1053-61. doi: 10.1002/ccd.21186. PMID 17525965
- [Background] Fukuda S, Gillinov AM, Liddicoat JR, Saracino G, Hayase M, Cohn WE, Schneider CW, Shiota T. Maintenance of geometric alterations associated with percutaneous mitral valve repair: real-time three-dimensional echocardiographic assessment in an ovine model. J Heart Valve Dis. 2008 May;17(3):276-82. PMID 18592924
- [Background] Daimon M, Gillinov AM, Liddicoat JR, Saracino G, Fukuda S, Koyama Y, Hayase M, Cohn WE, Ellis SG, Thomas JD, Shiota T. Dynamic change in mitral annular area and motion during percutaneous mitral annuloplasty for ischemic mitral regurgitation: preliminary animal study with real-time 3-dimensional echocardiography. J Am Soc Echocardiogr. 2007 Apr;20(4):381-8. doi: 10.1016/j.echo.2006.08.029. PMID 17400117
- [Background] Noble S, Bilodeau L. [Percutaneous therapies for aortic and mitral valvular disease]. Rev Med Suisse. 2007 May 30;3(113):1360-1, 1363-4, 1366-7. French. PMID 17645049
- [Background] Daimon M, Shiota T, Gillinov AM, Hayase M, Ruel M, Cohn WE, Blacker SJ, Liddicoat JR. Percutaneous mitral valve repair for chronic ischemic mitral regurgitation: a real-time three-dimensional echocardiographic study in an ovine model. Circulation. 2005 May 3;111(17):2183-9. doi: 10.1161/01.CIR.0000163547.03188.AC. Epub 2005 Apr 25. PMID 15851597
- [Background] Liddicoat JR, Mac Neill BD, Gillinov AM, Cohn WE, Chin CH, Prado AD, Pandian NG, Oesterle SN. Percutaneous mitral valve repair: a feasibility study in an ovine model of acute ischemic mitral regurgitation. Catheter Cardiovasc Interv. 2003 Nov;60(3):410-6. doi: 10.1002/ccd.10662. PMID 14571496